CLINICAL TRIAL: NCT06658977
Title: Open Label Rollover Study of Triumeq in Patients With Amyotrophic Lateral Sclerosis (ALS) Following the Lighthouse II Trial
Brief Title: RolloverTreatment With Triumeq for People With ALS Following the Lighthouse II Trial
Acronym: Lighthouse III
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This is a rollover study following the Lighthouse II trial; it was scheduled to stop when the LH II trial was stopped/completed. The LH II trial has been prematurely terminated so, likewise, this study has also now been stopped.
Sponsor: Macquarie University, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MQ2024003
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: Lighthouse
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — abacavir; Lamivudine; dolutegravir; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Intervention Model Description: Open Label Extension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triumeq open label (Experimental): Abacavir 600mg, Lamivudine 300mg and Dolutegravir 50mg ('Triumeq') one tablet daily
  Interventions: Drug: Abacavir 600mg, Lamivudine 300mg and Dolutegravir 50mg (Triumeq)

INTERVENTIONS:
Drug: Abacavir 600mg, Lamivudine 300mg and Dolutegravir 50mg (Triumeq) — One Triumeq tablet per day

SUMMARY:
Triumeq is an approved medicine for HIV. The effectiveness of Triumeq in Amyotrophic Lateral Sclerosis (ALS) is being investigated in the Lighthouse II trial. This study aims to assess whether Triumeq is safe and effective at delaying ALS disease progression when given long term. It is available for participants who have completed the Lighthouse II study. The main measurements are safety, tolerability and survival.

The study will go for approximately 2 years.

DETAILED DESCRIPTION:
Treatment options for ALS are very limited and there is a high unmet need for effective treatments. Triumeq targets a known neuron toxic pathway and is currently under investigation in a double blind placebo controlled trial, Lighthouse II. This study will be open to participants who took part in, and were still taking the study drug when they completed the Lighthouse II trial, in Australia and New Zealand.

The nature of the target and the mechanism of action of Triumeq are well understood. Participation in this rollover study is concurrent with standard of care, so participants are not limited in their use of therapies.

Participants will be assessed for adverse events, discontinuation of study medication, survival, measures of daily functioning, plus biomarker assessments of blood and urine samples.

Participant contacts may be face to face, or remote, and will be at 3 monthly intervals until approx December 2026 by which time it is anticipated the results of the Lighthouse II study will be available.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with ALS according to the Lighthouse II protocol who completed the Lighthouse II trial.
* Participants taking Riluzole must be on a stable dose.
* Participants taking taurursodiol supplements (TUDCA) can participate in this trial if the supplement does not contain sodium phenylbutyrate.
* Women must not become pregnant (e.g., post-menopausal, surgically sterile, using highly effective birth control methods or not having potentially reproductive sex) for the duration of the study plus five days; and women of childbearing potential must have a negative urine pregnancy test at baseline and be non-lactating.
* For participants taking antacids (regularly or as required), participant is willing and able to avoid taking antacids for at least 6 hours before and 2 hours after the Triumeq dose.
* Capable of providing informed consent and complying with the trial procedures.

Exclusion Criteria:

* In the Principal Investigator's opinion, the participant is unlikely to be compliant with the study drug dosing.
* People who are HLA-B*5701 positive.
* Presence of HIV antibodies at screening
* Presence of Hepatitis C antibodies at screening unless participants have had effective treatment for Hepatitis C
* Presence of Hepatitis B core or surface antigen at screening
* Known hypersensitivity to Dolutegravir, Abacavir or Lamivudine, or to any of the excipients.
* Moderate to severe hepatic impairment, as defined by local clinical guidelines.
* Participation in any other investigational drug trial or using another investigational drug within 5 half-lives of that drug.
* Use of NIV ≥22 h per day or having a tracheostomy
* Clinically significant history of unstable or severe cardiac, oncological, psychiatric, hepatic, or renal disease or other medically significant illness
* Taking medication contraindicated with Triumeq: Dofetilide or Fampridine (dalfampridine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | Duration of the study plus 7 days
  The primary endpoint of this trial is whether a patient had any drug related (definite, probable, possible) adverse events over the course of the extension trial. Tolerability is defined as the number of participants discontinuing study medication. Adverse events will be described in terms of relationship to temporary or permanent discontinuation of the study medication.

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Macquarie University, Neurology, North Ryde, New South Wales
  - Neuroscience Research Australia (NeuRA), Randwick, New South Wales
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, S.A.
  - Launceston General Hospital, Launceston, Tasmania
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - The Perron Institute, Nedlands, W.A.

IPD SHARING:
Plan to Share IPD: Yes
Contact Chief Investigator for access information
Supporting Information: Study Protocol
Access Criteria: Contact Chief Investigator for access information